CLINICAL TRIAL: NCT01980368
Title: Pilot Study of Effects of Tai Chi Easy on Cancer Survivors Experiencing Neuropathy
Brief Title: Tai Chi Easy in Treating Cancer Survivors With Peripheral Sensory Neuropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled-slow accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-007483; NCI-2016-01373 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-007483 (Other: Mayo Clinic in Arizona); P30CA015083 (NIH)
Record Dates: First submitted 2013-07-12; First posted 2013-11-11 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Cancer Survivor; Peripheral Sensory Neuropathy
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

ARMS (2):
- Group I (Tai Chi Easy) (Experimental): Patients attend Tai Chi Easy class for 60 minutes once a week for 6 weeks. Patients also receive a DVD and exercise manual of Tai Chi Easy exercises and are encouraged to practice at home for 30 minutes most days per week for 6 weeks.
  Interventions: Behavioral: Exercise Intervention; Other: Questionnaire Administration
- Group II (educational control) (Active Comparator): Patients receive readings each week and attend a book club to discuss the readings for 60 minutes once a week for 6 weeks.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive readings and attend book club
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group II (educational control)
Behavioral: Exercise Intervention — Receive Tai Chi Easy class, DVD, and exercise manual
  Arms: Group I (Tai Chi Easy)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well Tai Chi Easy works in treating cancer survivors with peripheral sensory neuropathy. Tai Chi Easy is a simple and repetitive form of exercise that consists of movements with meditation and may improve peripheral neuropathy symptoms among cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine effects of Tai Chi Easy (TCEasy) exercise intervention on peripheral sensory neuropathy of cancer survivors who have chemotherapy compared with an educational control (EC) intervention.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (TAI CHI EASY): Patients attend Tai Chi Easy class for 60 minutes once a week for 6 weeks. Patients also receive a DVD and exercise manual of Tai Chi Easy exercises and are encouraged to practice at home for 30 minutes most days per week for 6 weeks.

GROUP II (EDUCATIONAL CONTROL): Patients receive readings each week and attend a book club to discuss the readings for 60 minutes once a week for 6 weeks.

After completion of study, patients are followed up at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* 1 month - 5 years following completion of cytotoxic chemotherapy treatment for any cancer, and are experiencing neuropathy
* Self-report of >= 4 on the Peripheral Neuropathy Question

Exclusion Criteria:

* Recurrence of cancer or other active cancer
* Severe cachexia, dizziness, bone pain, or severe nausea (as judged by the investigator)
* Uncontrolled diabetes, untreated hypothyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
Change in peripheral sensory neuropathy, assessed by Peripheral Neuropathy Question, European Organization for Research and Treatment of Cancer (EORTC)-30, EORTC-Chemotherapy-induced peripheral neuropathy-20, and the modified Total Neuropathy Score | Baseline up to 2 months
  Will be assessed with a simple t-test of mTNS means. Additional analyses of factors assessed will similarly be conducted (and overall analysis of variance when combining outcome variable assessment at the three time points, and models of factor contribution with logistic regression if appropriate).

SECONDARY OUTCOMES:
Changes in anxiety assessed by POMS Total Mood Disturbance dimensions (tension-anxiety) | Baseline up to 2 months
Changes in body mass index assessed by weight and height | Baseline up to 2 months
  Will be measured directly using standardized protocols with medical-quality calibrated balance scales.
Changes in cognitive performance assessed by digit span and letter-number sequencing | Baseline up to 2 months
Changes in depression assessed by Program Operations Manual System (POMS) Total Mood Disturbance dimensions (depression-dejection) | Baseline up to 2 months
Changes in fatigue assessed by Fatigue Symptom Inventory | Baseline up to 2 months
Changes in pain assessed by Medical Outcomes Study-Short Form 36 | Baseline up to 2 months
Changes in sleep quality assessed by Pittsburgh Sleep Quality Index and actigraph | Baseline up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald Northfelt, Principal Investigator — Mayo Clinic